CLINICAL TRIAL: NCT00334529
Title: Evaluation of Alternative Oseltamivir (Tamiflu[R]) Dosing Strategies for Use During Influenza Prophylaxis
Brief Title: Alternative Oseltamivir Dosing Strategies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Richard T. Davey Jr., M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 060180; 06-I-0180
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-23

CONDITIONS: Influenza
Keywords: Tamiflu; Flu; Antiviral; Neuraminidase Inhibitor; Pharmacokinetic Trial; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir

SUMMARY:
This study will determine if oseltamivir (Tamiflu(Registered Trademark)) is safe and effective given less frequently than the currently prescribed dose of twice a day for 5 days to people who have the flu, and once a day for up to 6 weeks in people who have been exposed to someone else with flu and want to prevent getting it themselves. This study will see if the drug can be given once every other day instead of daily if given with another medication called probenecid (Benemid(Registered Trademark) or Probalan(Registered Trademark)).

Healthy people 18 years of age and older may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood and urine tests.

Participants are randomly assigned to one of the following regimens for 2 weeks: 1) 75 milligrams (mg) of oseltamivir once a day; 2) 75 mg of oseltamivir once every other day plus 500 mg probenecid four times a day; or 3) 75 mg of oseltamivir once every other day plus 500 mg probenecid twice a day. All medications are taken by mouth. On study day 0, subjects have the following baseline procedures: measurement of vital signs, review of medical and medication history, physical examination, blood draw and urine test. They also receive the first dose of oseltamivir or oseltamivir and probenecid. In addition, they undergo the following procedures as follows:

* Days 1 and 4: Vital signs; review of clinical symptoms, side effects and medications taken; urine testing and blood draw.
* Day 8: Same as day 1 plus count of study medication.
* Day 14: Same as day 8 plus pharmacokinetic study to measure the amount of oseltamivir and probenecid in the blood. For this test, a catheter is inserted into an arm vein and blood samples are collected through the catheter before taking the study medications, at the time the medications are taken, and again at 15 minutes, 30 minutes, 45 minutes and 1, 1.5, 2, 4, 8 and 12 hours after the medication is taken. The catheter is then removed. This is the last day to take the study medication.
* Day 15: Blood draw for 24-hour (post medication) blood sample.
* Day 16: Blood draw for 48-hour (post medication) blood sample.
* Days 21 and 28: Same as day 1.

DETAILED DESCRIPTION:
Pandemic influenza infection has the potential for causing significant morbidity and mortality in the United States and elsewhere. Oseltamivir (Tamiflu[R]) is a selective inhibitor of influenza virus neuraminidase and is U.S. FDA approved for both treatment and prophylaxis against influenza A and B viruses. However, at a time of national emergency, the supply of oseltamivir may be limited and alternative dosing strategies may be needed in order to provide as wide protection as possible from influenza or to treat as many infected patients as possible. Agents such as Probenecid that may extend the half-life of oseltamivir while maintaining effective oseltamivir plasma levels may potentially be useful in this regard. In this multi-center, three-arm, open-label, 48 patient trial, we propose to explore the relative safety and pharmacokinetics of oseltamivir plus Probenecid for 14 days in normal volunteers above and below the age of 65, according to the following dosing strategies: 16 subjects will be assigned to Group I Control Arm (Tamiflu[R] 75 mg given orally once daily), 16 subjects will be assigned to Group II Treatment Arm (Tamiflu [R] 75 mg orally once every other day plus Probenecid 500 mg orally four times daily), and 16 subjects will be assigned to Group III Treatment Arm (Tamiflu[R] 75 mg orally every other day and Probenecid 500 mg orally twice daily).

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will include males and non-pregnant females 18 years or older.

Subjects who can understand the study and potential safety concerns and can sign the informed consent form prior to admission to this study.

Subjects that are willing to complete all the required assessments, tests and evaluations and able to make all study visits.

1. Hemoglobin greater than or equal to 10.0 g/dL for males and greater than 9.0 g/dL for females;
2. Platelet count of greater than or equal to 75,000 /micro L;
3. Absolute neutrophil count greater than or equal to 1000 /micro L;
4. SGOT and SGPT less than 2.5 times normal upper limit;
5. Serum uric acid WNL;
6. Creatinine less than 1.5 times normal upper limit (normal UL 1.5 mg/dL) for the less than 65 years of age group and must be within normal limits for the greater than or equal to 65 years of age group;
7. creatinine clearance greater than or equal to 50 mL/min.

   EXCLUSION CRITERIA:

   Subjects with a creatinine clearance of less than 50 mL/min (as measured by the Cockcroft-Gault method)

   Subjects who are pregnant or breast feeding females

   Subjects who are not employing adequate contraception

   Subjects who are drug or alcohol abusers and in the opinion of the investigator would interfere with subject compliance and safety

   Subjects who are currently participating in any other clinical research study

   Any acute serious infection requiring prescription therapy within 14 days prior to Day 0 of the study

   Subjects with G6PD deficiency

   Subjects who may have been recently exposed to influenza

   Subjects with gout, blood dyscrasias, or history of hypersensitivity to sulfonamide drugs

   Subjects with contraindications to the study medications

   History of allergic reaction to probenecid

   Have kidney disease, kidney stones, or poorly functioning kidneys

   Have active peptic ulcer disease

   On high dose aspirin or any dose non-aspirin salicylate therapy

   Receiving any of the following medications (relative contraindication for probenecid):

   Acyclovir, allopurinol, penicillamine, clofibrate, rifampin, methotrexate, zidovudine, theophylline, dapsone, penicillins or cephalosporins, nonsteroidal anti-inflammatory drugs (NSAIDS) such as ibuprofen (Motrin, Advil, Nuprin, others), ketoprofen (Orudis, Oruvail, Orudis KT), diclofenac (Cataflam, Voltaren), etodolac (Lodine), fenoprofen (Nalfon), flurbiprofen (Ansaid), indomethacin (Indocin), ketorolac (Toradol), nabumetone (Relafen), oxaprozin (Daypro), piroxicam (Feldene), sulindac (Clinoril), tolmetin (Tolectin), and naproxen (Aleve, Anaprox, Naprosyn); a sulfa-based medication such as sulfamethoxazole (Bactrim, Septra, Gantanol), sulfasalazine (Azulfidine), sulfinpyrazone (Anturane), sulfisoxazole (Gantrisin), and others; an oral diabetes medicine such as glipizide (Glucotrol), glyburide (Micronase, Diabeta, Glynase), tolbutamide (Orinase), or tolazamide (Tolinase); a barbiturate such as phenobarbital (Luminal, Solfoton), amobarbital (Amytal), secobarbital (Seconal), and others; or a benzodiazepine (used to treat anxiety and panic disorders and to induce sleep) such as alprazolam (Xanax), diazepam (Valium), lorazepam (Ativan), temazepam (Restoril), chlordiazepoxide (Librium), clonazepam (Klonopin), clorazepate (Tranxene), oxazepam (Serax), estazolam (ProSom), flurazepam (Dalmane), quazepam (Doral), or triazolam (Halcion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2006-06-05; Primary Completion 2007-04-10 (Actual); Study Completion 2007-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Brooke Army Medical Center, Houston, Texas

REFERENCES:
- [Background] Osterholm MT. Preparing for the next pandemic. N Engl J Med. 2005 May 5;352(18):1839-42. doi: 10.1056/NEJMp058068. No abstract available. PMID 15872196
- [Background] Tumpey TM, Basler CF, Aguilar PV, Zeng H, Solorzano A, Swayne DE, Cox NJ, Katz JM, Taubenberger JK, Palese P, Garcia-Sastre A. Characterization of the reconstructed 1918 Spanish influenza pandemic virus. Science. 2005 Oct 7;310(5745):77-80. doi: 10.1126/science.1119392. PMID 16210530
- [Background] Taubenberger JK, Reid AH, Lourens RM, Wang R, Jin G, Fanning TG. Characterization of the 1918 influenza virus polymerase genes. Nature. 2005 Oct 6;437(7060):889-93. doi: 10.1038/nature04230. PMID 16208372